CLINICAL TRIAL: NCT05215665
Title: Efficacy, Safety Evaluation and Biomarker Screening of GEMOX Combined With Targeted Therapy and Immunotherapy for Patients With Advanced Cholangiocarcinoma
Brief Title: GEMOX Combined With Targeted Therapy and Immunotherapy for Patients With Advanced Cholangiocarcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GTIC
Record Dates: First submitted 2022-01-19; First posted 2022-01-31 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-05

CONDITIONS: Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — gemcitabine-oxaliplatin regimen; lenvatinib; toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Experimental): GEMOX+Lenvatinib+Toripalimab
  Interventions: Drug: GEMOX Regimen; Drug: Lenvatinib; Drug: Toripalimab
- group 2 (Experimental): GEMOX+Toripalimab
  Interventions: Drug: GEMOX Regimen; Drug: Toripalimab

INTERVENTIONS:
Drug: GEMOX Regimen — Oxaliplatin 100mg/m2 IV d1 Q3W+ gemcitabine 1000mg/m2 IV d1/8 Q3W
Drug: Lenvatinib — 8/12mg PO QD continuously
  Arms: group 1
Drug: Toripalimab — 240mg IV d1 Q3W

SUMMARY:
The clinical trial is designed to evaluate the safety and efficacy of GEMOX combined with targeted therapy and immunotherapy for patients with advanced cholangiocarcinoma, and screen the potential biomarkers

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years old ≤ age ≤ 70 years old
* ECOG PS scores 0-1
* Expected survival time > 12 weeks
* Advanced cholangiocarcinoma confirmed by histopathology and/or cytology, locally advanced (inoperable) or distant metastasis, and with at least one measurable lesion that has not been locally treated (per RECIST 1.1 criteria)
* Not received any previous systemic or local treatment for the tumor
* Sufficient organ and bone marrow function

Exclusion Criteria:

* Suffered from other malignant tumors in the past 5 years (except Radical basal cell carcinoma of the skin squamous carcinoma of the skin and/or radical resected carcinoma in situ)
* Ampullary tumor
* Received treatment from other clinical trials within 4 weeks before the first dose
* Received any anti-PD-1 antibody, anti-PD-L1/L2 antibody, anti-CTLA4 antibody, or other immunotherapy
* Suffered from severe cardiovascular disease within 12 months before enrollment, such as symptomatic coronary heart disease, congestive heart failure ≥ Grade II, uncontrolled arrhythmia, and myocardial infarction
* Uncontrollable pleural effusion, pericardial effusion or ascites
* Use steroids or other systemic immunosuppressive therapies 4 weeks before enrollment
* Allergic reactions to the drugs used in this study
* HIV antibody positive, active hepatitis B or C (HBV, HCV)
* Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation
* other conditions that the investigator deems inappropriate for enrollment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | up to 90 days after last treatment administration
  Overall response rate ( ORR) is defined as proportion of participants who have a best response of CR or PR

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | up to 90 days after last treatment administration
  Disease Control Rate (DCR) is defined as proportion of participants who have a best response of CR、PR or SD
Progression free survival (PFS) | up to 3 years
  the time period from randomization of the participants to objective tumor progression or death
Overall survival (OS) | up to 3 years
  the time period from the randomization of the participants to the death event due to any reason
The frequency, duration, and severity of adverse events | up to 30 days after last treatment administration
  Safety is assessed by the frequency, duration, and severity of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality, China